CLINICAL TRIAL: NCT03564951
Title: Comparison of Ablation of Anisochronous Zones vs Spatio-temporal Dispersal Zones in Addition to Antral Electrical Isolation During Radiofrequency Treatment of Paroxysmal or Persistent Atrial Fibrillation
Brief Title: Ablation of Anisochronous Zones vs Spatio-temporal Dispersal Zones With Antral Electrical Isolation During Radiofrequency Treatment of Paroxysmal or Persistent Atrial Fibrillation
Acronym: ISOCHRONE-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIMAO/2017-02/MG-01
Record Dates: First submitted 2018-06-11; First posted 2018-06-21 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): ablation of Atrial fibrillation using spatio-temporal dispersion
  Interventions: Procedure: Atrial fibrillation ablation
- Isochrone (Experimental): ablation of concordance zones using isochrone and voltage maps
  Interventions: Procedure: Atrial fibrillation ablation

INTERVENTIONS:
Procedure: Atrial fibrillation ablation — ablation of Atrial fibrillation using spatio-temporal dispersion
  Arms: Control
Procedure: Atrial fibrillation ablation — ablation of concordance zones using isochrone and voltage maps
  Arms: Isochrone

SUMMARY:
Using isochronous maps during radiofrequency ablation procedures may identify the driver zones responsible for atrial fibrillation maintenance with greater accuracy compared to a conventional procedure (simple antral isolation of the associated pulmonary veins or, if necessary, combined with removal of spatio-temporal dispersal zones) that do not use isochronous maps, and thus improve the efficiency and safety of atrial fibrillation treatment by radiofrequency treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* The patient is at least 18 years old
* The patient has paroxysmal or persistent atrial fibrillation
* The patient is available for 18 month follow-up

Exclusion Criteria:

* The subject is participating in a category 1 interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* The patient is pregnant or breastfeeding
* Sinus rhythm has not been able to be determined using external electric cardioversion
* Patient not susceptible to atrial fibrillation following wide antrum circle ablation
* The subject has already been included in the study (patients cannot be included more than once)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2020-08-19 (Actual); Study Completion 2020-08-19 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation relapse between groups | Month 18
  Atrial fibrillation detected by routine or event-associated Holter examination

SECONDARY OUTCOMES:
Atrial fibrillation relapse between groups | Month 12
  Atrial fibrillation detected by routine or event-associated Holter examination
Arrhythmia occurrence between groups | Month 12
  Arrhythmia, including atrial tachycardia detected by routine or event-associated Holter examination
Arrhythmia occurrence between groups | Month 18
  Arrhythmia, including atrial tachycardia detected by routine or event-associated Holter examination
Concordance of isochrone and voltage maps | Day 0
  Binary yes/no
Maximum variation of conduction speed between variation healthy zones with anisochronic zones in the same anatomic region | Day 0
Comparison of the decreasing velocities between healthy zones and anisochronic zones in the same anatomic region | Day 0
Comparison of wave front rotation between healthy zones and anisochronic zones in the same anatomic region | Day 0
  degrees
Total time of radiofrequency between groups | Day 0
  Minutes
Comparison of lesion volume between groups | Day 0
  Force-time integral, lesion size index or stroke volume index
Total procedure time between groups | Day 0
  Minutes
Number of treated zones between groups | Day 0
Size of treated zones between groups | Day 0
  cm2
List locations most frequently treated | Day 0
  Number of each
Survival without relapse of the subgroups paroxysmal versus persistent atrial fibrillation. | Month 18
  Atrial fibrillation detected by routine or event-associated Holter examination
Survival without relapse of the subgroups treated using the Carto- vs Rhythmia-guided ablation approaches. | Month 18
  Atrial fibrillation detected by routine or event-associated Holter examination

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Montpellier, Montpellier
  - CHU Nimes, Nîmes